CLINICAL TRIAL: NCT02364973
Title: Combined PET-MRI in the Diagnostics of Chronic Inflammatory Bowel Diseases (IBD)- a Feasibility Study
Status: Completed | Type: Observational
Sponsor: Turku University Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: T31/2014
Record Dates: First submitted 2014-12-03; First posted 2015-02-18 (Estimated); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: IBD

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- PET-MRI: Patients with chronic inflammatory bowel disease who are treated at Turku University hospital outpatient clinic or ward
  Interventions: Other: PET-MRI

INTERVENTIONS:
Other: PET-MRI — The study patients undergo positron emission tomography (PET) after informed consent is obtained

SUMMARY:
The main purpose of the present study is to examine the diagnostic performance of combined PET-MRI in detecting colonic and small bowel wall inflammatory processes caused by ulcerative colitis and Crohn's disease.

DETAILED DESCRIPTION:
COMBINED PET-MRI IN THE DIAGNOSTICS OF CHRONIC INFLAMMATORY BOWEL DISEASES (IBD)- A FEASIBILITY STUDY (RESEARCH CODE T31/2014)

1. Background

   Ulcerative colitis and Crohn's disease are chronic inflammatory bowel diseases (IBD) with relapsing and remitting course. The incidence of IBD is highest in teenagers and young adults, but IBD may also affect children and old people. The diagnosis of IBD is based on clinical symptoms, endoscopy and histology of the bowel wall.

   Aims of the study

   The main purpose of the present study is to examine the diagnostic performance of combined PET-MRI in detecting colonic and small bowel wall inflammatory processes caused by ulcerative colitis and Crohn's disease.

   The hypothesis of the study is a) IBD-related inflammatory changes are detected by PET-MRI (18 F-FDG) and correlate with the endoscopic and histologic activity of colitis and ileitis.

   Study design

   A total of 45 IBD patients (ulcerative colitis or Crohn's disease) aged over 15 years will be recruited from the patients visiting outpatient gastroenterology clinic of Turku University Hospital. Every patient undergoes colonoscopy with biopsy specimens, endoscopic and histologic data are recorded via structured forms. Laboratory specimens with samples for biobank are obtained. Then the patients are examined by abdominal MRI and PET.

   Inclusion criteria:
   * informed consent obtained
   * age over 18 years
   * diagnosis of ulcerative colitis or Crohn's colitis based on endoscopy and histology
   * the activity of colitis confirmed by histology and/or elevated fecal calprotectin concentration
   * fertile women have contraception
   * no previous abdominal surgery
   * no X-ray investtigations during preceding year
2. Investigators

   Principal investigator Markku Voutilainen, MD, Department of Gastroenterology

   Other investigators Hannu Aronen, Sami Kajander, Johanna Virtanen, Virva Saunavaara, Department of Radiology and PET center.

   Mervi Tenhami, Saila Kauhanen, Department of surgery

   Pirjo Nuutila, Department of Endocrinology and PET center

   Jukka Kemppainen, physicist, PET center

   Olli Carpen, Department of pathology

   Ville Aalto, statistician, University of Turku,
3. PET tracer is 18 F-FDG, dose 280 megabequerel (MBq, bowel imaging)
4. Data of scans and details of scanning time (including positioning and transmission) by tracer, blood sampling (activity, metabolites)

   * Before scanning: oral contrast intake (Mannitol dilution) 65 min
   * Magnetic resonance imaging (MRI) positioning (prone position) 5min
   * Abdominal MRI Scanning: 50min
   * Region: from diaphragma to symphysis
   * During the scan: i.v. Buscopan and +Gadolinium
   * Sequences (fast gradient echo, predominantly breath-hold imaging):

     1. T2 (field echo type) cor and ax
     2. T2
     3. T1 fs cor and ax +Gd
     4. T1 fs repeated (start at 40 seconds after injection)
     5. Diffusion
     6. T2 or T1 cor +aks
   * PET, FDG tracer: 15 min

     * Total scanning time including positioning, MRI and PET: 70 min

   Scanning code JN5JS (= Large scale PET-MRI of the body)
5. Number of study subjects 45
6. Scanner PET/MRI
7. The radiation dose will be calculated by physicist after the tracer, it's amount and detector are determined. The permission from ethical committee was obtained in August 2014..
8. No quality issues (QA), routine radiological quality control
9. The study has been accepted by the Ethical committee of Turku University Hospital
10. Present study is academic study and all data relating to the study belongs to the investigators.
11. The test patients are to undergo the study in September 2014. The study is to be started October 2014.
12. For the financing of the study, VTR-/EVO-funding (Funding from the Finnish government) will be applied. At present, 6000€ have been obtained from research funding of Department of internal medicine.

ELIGIBILITY:
Inclusion Criteria

* age over 18 years
* IBD (ulcerative colitis or Crohn's disease diagnosed by endoscopy and/or radiology
* no previous abdominal surgery
* no biological therapy for IBD

Exclusion Criteria:

* pregnancy
* diabetes
* the patient is unable to give informed consent

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: IBD patients living in the Turku University Hospital referral area
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2014-11 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2020-08 (Actual)

PRIMARY OUTCOMES:
The percentage of patients with active inflammation detected by PET-MRI | 3 YEARS
  COMBINED PET-MRI IN THE DIAGNOSTICS AND FOLLOW-UP OF CHRONIC INFLAMMATORY BOWEL DISEASES

CONTACTS AND LOCATIONS:
Overall Officials: Markku Voutilainen, MD, Principal Investigator — Turku University Hospital
Locations (1):
- Turku University Hospital, Turku, Finland